CLINICAL TRIAL: NCT05303116
Title: COVID19 Effects on the Brain and Cerebral Function; Do Quantitative Measures of Brain Electrical Activity Along With Neurocognitive Assessments Correlate With Symptoms and Clinical Assessment?
Brief Title: Do EEG and Neurocognitive Assessments Correlate With COVID Brainfog Symptoms?
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Collaborators: BrainScope Company, Inc. (Industry)
Responsible Party: Principal Investigator, Edward Michelson, MD, Professor and Chair, Dept of Emergency Medicine, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: E22060
Record Dates: First submitted 2022-03-28; First posted 2022-03-31 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
Keywords: COVID-19; "brain fog"; altered mental status
MeSH Terms: conditions — COVID-19; Mental Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control: Patients with COVID who are NOT experiencing altered mental status
  Interventions: Diagnostic Test: Brainscope modified EEG and cognitive testing
- COVID patients: COVID patients who are experiencing confusion,
  Interventions: Diagnostic Test: Brainscope modified EEG and cognitive testing

INTERVENTIONS:
Diagnostic Test: Brainscope modified EEG and cognitive testing — Modified EEG performed using BrainScope device along with cognitive testing performed with BrainScope device and other surveys.

SUMMARY:
Since the neurologic symptoms of some COVID patients ('brain fog') resemble those of patients with concussion, the aim of this study is to identify EEG and cognitive function changes in COVID patients. We will use the FDA cleared BrainScope medical device in conjunction with standard neurocognitive tests to identify correlations with electrical biomarkers and to potentially identify new, unique patterns of altered brain electrical activity associated with COVID-19 infection. A baseline assessment will be performed shortly after hospital presentation and then a second evaluation will be performed 45-60 days post hospital discharge to reassess clinical status, brain electrical biomarkers and neurocognitive performance. The goal will be to develop an objective measurement of brain function/dysfunction associated with COVID-19 infection which might be employed in future studies of treatments for COVID-19 brain fog and to aid in tracking recovery.

DETAILED DESCRIPTION:
1. Screening and Consent - Patients with a diagnosis of COVID-19 will be asked by the research personnel if they are experiencing symptoms of 'brain fog' (confusion, altered memory, headache, trouble concentrating.) Those responding affirmatively will be asked to complete a brief mental status exam (mini MoCA). Those patients scoring 25 or less out of 30 will then move forward to the formal written consent process. We will also recruit 5 control patients who are COVID positive but are not experiencing 'brainfog' symptoms.
2. Electroencephalogram (EEG) - We will perform an EEG using a Brainscope device.
3. Neurocognitive Assessment (brain function tests) - While the EEG electrodes are still attached, we will perform these assessments that test attention, concentration, reaction time, processing speed, decision making, and executive function. These are called the Structural Injury classifier (SIC) and Concussion Index (CI) assessments that are computed using FDA cleared algorithms for the likelihood of structural brain injury and the likelihood and severity of brain function impairment.
4. Full MoCA assessment - After the Brainscope evaluation patients will be asked questions on the paper-based full MoCA cognitive assessment and the score will be recorded.
5. Concussion Symptom Inventory (CSI) - Study personnel will ask questions about symptoms using the CSI which is a standardized tool for evaluating injured patients who have concussion.
6. Inventory of COVID Symptoms - Research personnel will collect information about COVID symptoms using standardized PROMIS surveys. (Dyspnea severity and Physical Function)
7. Demographics - We will collect demographic information that includes age and sex, along with vital signs, pulse oximetry, and supplemental oxygen requirement, physical exam, neurological exam, lab test results, medications given during hospitalization, and results of any imaging done on the head during hospitalization. Standard laboratory results including blood counts, chemistry and biomarkers of inflammation obtained as standard of care will be recorded.
8. Follow-up Visit - Participants will return to the clinic for a follow-up visit 45-60 days after discharge from the hospital. At that visit the Brainscope EEG, mental function tests, and symptom surveys will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Current COVID 19 infection
* Experiencing 'brain fog' symptoms (e.g.confusion, mental slowness, unable to concentrate)
* GCS of 14 or 15
* sufficient mental capacity to provide informed consent
* hemodynamically stable
* able to cooperate with EEG collection and neurometric testing
* admitted to a floor bed rather than ICU

Exclusion Criteria:

* Head or facial trauma
* Any abnormality that would prevent electrodes from being placed on the head
* Known central nervous system (CNS) disease i.e. MS, Parkinson's disease
* Know seizure disorder
* Known dementia
* Metabolic encephalopathy i.e. uremia, hepatic
* Alcohol intoxication to the point they cannot give consent
* Hypoxia that is not corrected to 92% by nasal cannula, or simple face mask
* Chronic alcohol or drug dependence
* Prior cerebrovascular accident (CVA)
* Prior brain surgery
* Known brain mass
* Receiving sedation medications at time of consent
* End stage renal disease (ESRD) on dialysis
* Acute psychosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with COVID-19 infection who are experiencing 'brain fog' symptoms and who will admitted to the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Identify unique brain electrical activity in patients who have COVID-19 infection and 'brain fog' symptoms | Baseline and follow-up evaluations (45-60 days after hospital discharge)
  Compile types of EEG changes demonstrated by COVID patients with 'brain fog' symptoms compared to COVID patients without 'brain fog' symptoms.

SECONDARY OUTCOMES:
Persistence of neurocoginitive dysfunction over time | Baseline and follow-up evaluations (45-60 days after hospital discharge)
  Comparison of neurocognitive test results at baseline and follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Edward Michelson, MD, Principal Investigator — Chair, Dept of Emergency Medicine; TTUHSC El Paso
Locations (1):
- University Medical Center of El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maury A, Lyoubi A, Peiffer-Smadja N, de Broucker T, Meppiel E. Neurological manifestations associated with SARS-CoV-2 and other coronaviruses: A narrative review for clinicians. Rev Neurol (Paris). 2021 Jan-Feb;177(1-2):51-64. doi: 10.1016/j.neurol.2020.10.001. Epub 2020 Dec 16. PMID 33446327
- [Background] Graham EL, Clark JR, Orban ZS, Lim PH, Szymanski AL, Taylor C, DiBiase RM, Jia DT, Balabanov R, Ho SU, Batra A, Liotta EM, Koralnik IJ. Persistent neurologic symptoms and cognitive dysfunction in non-hospitalized Covid-19 "long haulers". Ann Clin Transl Neurol. 2021 May;8(5):1073-1085. doi: 10.1002/acn3.51350. Epub 2021 Mar 30. PMID 33755344
- [Background] Lambrecq V, Hanin A, Munoz-Musat E, Chougar L, Gassama S, Delorme C, Cousyn L, Borden A, Damiano M, Frazzini V, Huberfeld G, Landgraf F, Nguyen-Michel VH, Pichit P, Sangare A, Chavez M, Morelot-Panzini C, Morawiec E, Raux M, Luyt CE, Rufat P, Galanaud D, Corvol JC, Lubetzki C, Rohaut B, Demeret S, Pyatigorskaya N, Naccache L, Navarro V; Cohort COVID-19 Neurosciences (CoCo Neurosciences) Study Group. Association of Clinical, Biological, and Brain Magnetic Resonance Imaging Findings With Electroencephalographic Findings for Patients With COVID-19. JAMA Netw Open. 2021 Mar 1;4(3):e211489. doi: 10.1001/jamanetworkopen.2021.1489. PMID 33720371
- [Background] Bazarian JJ, Elbin RJ, Casa DJ, Hotz GA, Neville C, Lopez RM, Schnyer DM, Yeargin S, Covassin T. Validation of a Machine Learning Brain Electrical Activity-Based Index to Aid in Diagnosing Concussion Among Athletes. JAMA Netw Open. 2021 Feb 1;4(2):e2037349. doi: 10.1001/jamanetworkopen.2020.37349. PMID 33587137
- [Background] Hanley D, Prichep LS, Bazarian J, Huff JS, Naunheim R, Garrett J, Jones EB, Wright DW, O'Neill J, Badjatia N, Gandhi D, Curley KC, Chiacchierini R, O'Neil B, Hack DC. Emergency Department Triage of Traumatic Head Injury Using a Brain Electrical Activity Biomarker: A Multisite Prospective Observational Validation Trial. Acad Emerg Med. 2017 May;24(5):617-627. doi: 10.1111/acem.13175. Epub 2017 Mar 31. PMID 28177169
- [Background] Hanley D, Prichep LS, Badjatia N, Bazarian J, Chiacchierini R, Curley KC, Garrett J, Jones E, Naunheim R, O'Neil B, O'Neill J, Wright DW, Huff JS. A Brain Electrical Activity Electroencephalographic-Based Biomarker of Functional Impairment in Traumatic Brain Injury: A Multi-Site Validation Trial. J Neurotrauma. 2018 Jan 1;35(1):41-47. doi: 10.1089/neu.2017.5004. Epub 2017 Sep 21. PMID 28599608